CLINICAL TRIAL: NCT04548115
Title: ARTISAN 2.0: Deconstructing the Integrative Efficacy of a Multimodal Art-based Intervention to Strengthen Understanding and Demystify Misconceptions on Arts, Heritage, and Health
Brief Title: ARTISAN 2.0: Deconstructing the Integrative Efficacy of a Multimodal Art-based Intervention
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Nanyang Technological University (Other)
Collaborators: National Museum of Singapore (Unknown)
Responsible Party: Principal Investigator, Andy Hau Yan Ho, PhD, EdD, Associate Professor, Nanyang Technological University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: IRB-2020-02-006
Record Dates: First submitted 2020-09-09; First posted 2020-09-14 (Actual); Last update posted 2020-09-14 (Actual); Status verified 2020-09

CONDITIONS: Intergenerational Relations; Loneliness; Well Aging
Keywords: Arts-based Intervention, Cultural Heritage

STUDY DESIGN:
Intervention Model Description: Using site randomization, each higher education institution will be randomized into one of the five RCT conditions (i.e. full ARTISAN, participatory arts, art space, storytelling and control), and each elderly care agency will be randomized into one of the same five conditions. Based on randomization outcome, one higher education institution will be paired with one elderly care agency, the paired collaborating sites will be allocated to the same RCT condition. Participant recruitment will be simultaneously conducted at each paired sites through 5 sequential rounds, and each round will recruit 2 groups, totalling 10 groups for the entire study. Each group will comprise 14 participants with youths and senior to be randomized paired as dyads, who will undergo a 5-week RCT condition with a follow-up assessment at 10-weeks. At any given time during the study, 2 groups will be run concurrently until all 10 groups complete the RCT.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (5):
- ARTISAN Condition (Experimental): Participants assigned to this arm will engage in ARTISAN, a 5-weekly, 15-hour group-based arts and heritage intervention programme with specific intervention components including curated museum tours, facilitated storytelling and professionally-led art-making. The weekly intervention covers the five ARTISAN themes of national heritage, social bonds, adversity and resilience, dreams and aspiration, and community art exhibition.
  Interventions: Behavioral: ARTISAN Condition
- Intergenerational Participatory Arts Condition (Experimental): Participants assigned to this arm will engage in the participatory arts-making component of the ARTISAN Intervention framework. Youths and senior participants in this condition will engage in a 5-weekly, 5-hour, group-based professionally-led art-making that covers the five ARTISAN themes.
  Interventions: Behavioral: Intergenerational Participatory Arts Condition
- Intergenerational Art-space Condition (Experimental): Participants assigned to this arm will engage in the cultural space component of the ARTISAN Intervention framework. Youths and senior participants in this condition will engage in a 5-weekly, 5-hour, group-based a group-based curated museum tour that covers the five ARTISAN themes.
  Interventions: Behavioral: Intergenerational Art-space Condition
- Inter-generational Storytelling Condition (Experimental): Participants assigned to this arm will engage in the storytelling component of the ARTISAN Intervention framework. Youths and senior participants in this condition will be paired to engage in a 5-weekly, 5-hour, group-based guided storytelling activity that covers the five ARTISAN themes.
  Interventions: Behavioral: Intergenerational Storytelling Condition
- Control Condition (Experimental): Participants assigned to this arm will engage in a 5-weekly, 5-hour, group-based physical activity session conducted in the community.
  Interventions: Behavioral: Control Condition

INTERVENTIONS:
Behavioral: ARTISAN Condition — Youth and senior participants will be randomly paired and engage in the 5-weekly, 3-hour ARTISAN intervention as dyads (totaling 15 hours of intervention). In the first four weeks of the ARTISAN, dyads will engage in themed museum tours facilitated by a docent (45min), guided storytelling (45 min) and professionally-led art-making (45 min). The remaining time (45 min) is allocated for session breaks, session introduction/closing, and buffer time for movement around the gallery. The final week involves an exhibition where participants share their artworks with the public and reflect on their experiences and artworks. The weekly session themes are as follows: Week 1: Discovering our National Heritage (Art medium: Clay); Week 2: Strengthening Social Bonds (Art medium: Acrylic Paints); Week 3: Overcoming Adversities and Resilience (Art medium: Beads); Week 4: Building Dreams and Aspirations (Art medium: Recycled Materials); Week 5: Sharing our Stories and Legacies (Community Showcase)
  Arms: ARTISAN Condition
Behavioral: Intergenerational Participatory Arts Condition — Youths and senior participants in this condition will be randomly paired and engage in a 5-weekly 45-minute group-based art activity conducted in a community space with 15 minutes of preparation/break time (totaling 5 hours of intervention). A professional artist or art therapist will facilitate art-making sessions with the participants in a community space, utilizing the same mediums that were used in ARTISAN. The weekly session themes are as follows: Week 1: Discovering our National Heritage (Art medium: Clay); Week 2: Strengthening Social Bonds (Art medium: Acrylic Paints); Week 3: Overcoming Adversities and Resilience (Art medium: Beads); Week 4: Building Dreams and Aspirations (Art medium: Recycled Materials); Week 5: Sharing our Stories and Legacies (Community Showcase)
  Arms: Intergenerational Participatory Arts Condition
Behavioral: Intergenerational Art-space Condition — Youths and senior participants in this condition will engage in a 5-weekly 45-minute group-based curated museum tour that follow the ARTISAN themes with 15 minutes of preparation/break time, and conducted by a trained docent at the National Museum Singapore (totaling 5 hours of intervention).The weekly session themes are as follows: Week 1: Discovering our National Heritage; Week 2: Strengthening Social Bonds; Week 3: Overcoming Adversities and Resilience; Week 4: Building Dreams and Aspirations; Week 5: Sharing our Stories and Legacies.
  Arms: Intergenerational Art-space Condition
Behavioral: Intergenerational Storytelling Condition — Youths and senior participants in this condition will be paired to engage in a 5-weekly 45 minute group-based storytelling activity conducted in a community space with 15 minutes of preparation/break time (totaling 5 hours of intervention). Storytelling sessions will be conducted by a trained facilitator, and conversation starters from ARTISAN intervention will be used. The weekly session themes are as follows: Week 1: Discovering our National Heritage; Week 2: Strengthening Social Bonds; Week 3: Overcoming Adversities and Resilience; Week 4: Building Dreams and Aspirations; Week 5: Sharing our Stories and Legacies.
  Arms: Inter-generational Storytelling Condition
Behavioral: Control Condition — Participants in this condition will engage in a 5-weekly 45 minute group-based physical activity session conducted in the community with 15 minutes of preparation/break time (totaling 5 hours of intervention). Physical activity was selected over basic psychosocial care to test the effects of inter-generational contact independent of arts and heritage-based engagements.
  Arms: Control Condition

SUMMARY:
To address perceived loneliness via citizen empowerment, ARTISAN (Aspiration and Resilience Through Intergenerational Storytelling and Art-based Narratives) was developed by the Principal Investigator in partnership with the National Arts Council and the National Museum of Singapore. A 2018 pilot study was conducted with the aim to establish ARTISAN's intervention framework, as well as to evaluate the effectiveness of the intervention in promoting resilience, social connectedness, wellbeing, personhood and nationhood. The current research builds on the empirical foundation of the pilot study and seeks to deconstruct the ARTISAN intervention for gaining a deeper understanding of its underlying mechanisms for promoting positive life changes among youth and senior participants such as reduced loneliness, enhanced resilience, psychological wellbeing, social connectedness and sense of nationhood.

DETAILED DESCRIPTION:
Objective: The core objective is to critically investigate and assess the independent and combined efficacy of each key intervention components of ARTISAN's multimodal framework, which consist of: 1) full ARTISAN condition; 2) intergenerational participatory arts condition; 3) intergenerational art space condition; 4) intergenerational storytelling condition; and 5) control condition of physical activity.

Methods: Utilizing a five-arm, multicentre randomized controlled trial (RCT) design, 70 youths and 70 seniors (N=140) from 10 collaborating sites will be invited to participate in a 5-weeks intervention programme under one of five conditions (ARTISAN condition, Participatory Arts condition, Art-space condition, Storytelling condition, Control condition). Quantitative measurements will be taken at baseline, immediately after the intervention, and ten week post baseline the interventions.

Significance: The results generated will serve to illuminate the intricate pathways in which arts and heritage can cultivate positive life changes, and address misconceptions and about the pivotal roles that arts and heritage play in health promotion.

ELIGIBILITY:
Inclusion Criteria:

* Youth between the age of 16 to 35
* Community-dwelling seniors above the age of 60
* Fluent in verbal English or Mandarin

Exclusion Criteria:

* Individuals who are unable to provide informed consent (or parental consent where applicable)
* Individuals diagnosed with major mental illness or cognitive impairment (If deemed appropriate, potential senior participants will be screened by the NTU research team using the Mini-Mental State Examination (MMSE))
* Participants who had engaged in the ARTISAN pilot study

Min Age: 16 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 140 (Estimated)
Dates: Start 2020-12 (Estimated); Primary Completion 2022-11 (Estimated); Study Completion 2022-11 (Estimated)

PRIMARY OUTCOMES:
Change in Loneliness (ULS-8) scores from baseline | Participants will be assessed at three time points: [T1] baseline; [T2] immediately post-intervention/second baseline (5 weeks post T1); and [T3] 5 weeks follow-up/ immediately post-intervention (5 weeks post T2).
  The 8-item UCLA Loneliness Scale (ULS-8) is used to assess Loneliness. Participants will be asked to indicate their agreement for statements on a 4-point scale.
Changes in Resilience (ER-11) scores from baseline | Participants will be assessed at three time points: [T1] baseline; [T2] immediately post-intervention/second baseline (5 weeks post T1); and [T3] 5 weeks follow-up/ immediately post-intervention (5 weeks post T2).
  Resilience is assessed by the 11-item refined version of Ego-Resilience Scale (ER-11). Participants will be asked to indicate their agreement for statements on a 4-point scale.
Changes in Social Connectedness (MOS-SS) scores from baseline | Participants will be assessed at three time points: [T1] baseline; [T2] immediately post-intervention/second baseline (5 weeks post T1); and [T3] 5 weeks follow-up/ immediately post-intervention (5 weeks post T2).
  Social Connectedness is measured by the Emotional, Affectionate, and Positive Interaction sub-scales of the Medical Outcome Study Social Support Survey (MOS-SS). Participants will be asked to respond to 14-items on a 5-point likert scale.
Changes in National and Cultural Identity (NATID) scores from baseline | Participants will be assessed at three time points: [T1] baseline; [T2] immediately post-intervention/second baseline (5 weeks post T1); and [T3] 5 weeks follow-up/ immediately post-intervention (5 weeks post T2).
  National identity is assessed by a modified version of the National Identity Scale (NATID) which comprises 8-items. Participants will be asked to rate their agreement on statements regarding national heritage and cultural homogeneity on a 7-point likert scale.

SECONDARY OUTCOMES:
Changes in Psychological wellbeing (PWB) scores from baseline | Participants will be assessed at three time points: [T1] baseline; [T2] immediately post-intervention/second baseline (5 weeks post T1); and [T3] 5 weeks follow-up/ immediately post-intervention (5 weeks post T2).
  Psychological wellbeing is measured by the Personal Growth and Self-Acceptance sub-scales of the Ryff's Psychological Wellbeing Scale (PWB) which comprises 18 items.
Changes in Depressive symptoms (PHQ-4) scores from baseline | Participants will be assessed at three time points: [T1] baseline; [T2] immediately post-intervention/second baseline (5 weeks post T1); and [T3] 5 weeks follow-up/ immediately post-intervention (5 weeks post T2).
  Depressive symptoms is assessed by the 4-item brief version of the Patient Health Questionnaire (PHQ-4).
Changes in Self-esteem (RSES-4) scores from baseline | Participants will be assessed at three time points: [T1] baseline; [T2] immediately post-intervention/second baseline (5 weeks post T1); and [T3] 5 weeks follow-up/ immediately post-intervention (5 weeks post T2).
  Self-esteem is measured by the 4-item shortened-version of the Rosenberg's Self-Esteem Scale (RSES-4).
Changes in Life satisfaction (SWLS) scores from baseline | Participants will be assessed at three time points: [T1] baseline; [T2] immediately post-intervention/second baseline (5 weeks post T1); and [T3] 5 weeks follow-up/ immediately post-intervention (5 weeks post T2).
  Life satisfaction is assessed by the single-item Satisfaction with Life Scale (SWLS).
Changes in Quality of life (WHOQoL-8) scores from baseline | Participants will be assessed at three time points: [T1] baseline; [T2] immediately post-intervention/second baseline (5 weeks post T1); and [T3] 5 weeks follow-up/ immediately post-intervention (5 weeks post T2).
  Perceived quality of life is measured by the 8-item WHO Quality of Life Scale-8 (WHOQoL-8/EUROHIS-QOL).
Changes in Spiritual wellbeing (FACIT-Sp) scores from baseline | Participants will be assessed at three time points: [T1] baseline; [T2] immediately post-intervention/second baseline (5 weeks post T1); and [T3] 5 weeks follow-up/ immediately post-intervention (5 weeks post T2).
  Spiritual wellbeing is measured by the 8-item peace and meaning subscales of the Functional Assessment of Chronic Illness Therapy - Spiritual Well-Being Scale (FACIT-Sp).

CONTACTS AND LOCATIONS:
Overall Officials: Andy HY Ho, PhD, EdD, Principal Investigator — Nanyang Technological University
Locations (1):
- Nanyang Technological University, Singapore, Singapore

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- See also: ARTISAN Pilot Study Introduction — https://blogs.ntu.edu.sg/arch/2018/07/27/artisan/